CLINICAL TRIAL: NCT02327299
Title: Assessment of the Bioavailability of Iron in Iron Fortified Bouillon Cubes in Healthy Women
Brief Title: Iron Bioavailability From Cubes
Acronym: Fe Bouillon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FDS-SAV-1615
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Iron Deficiency
Keywords: Iron deficiency; Iron fortification
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FePP (Experimental): Bouillon fortified with 4mg FePP
  Interventions: Dietary Supplement: Bouillon fortified with FePP
- FePP + Stabilizer (Experimental): Bouillon fortified with 4mg FePP + Stabilizer
  Interventions: Dietary Supplement: Bouillon fortified with FePP + Stabilizer
- FeSO4 (Experimental): Bouillon fortified with 4mg FeSO4
  Interventions: Dietary Supplement: Bouillon fortified with FeSO4
- FeSO4 + Stabilizer (Experimental): Bouillon fortified with 4mg FeSO4 + Stabilizer
  Interventions: Dietary Supplement: Bouillon fortified with FeSO4 + Stabilizer

INTERVENTIONS:
Dietary Supplement: Bouillon fortified with FePP
  Arms: FePP
Dietary Supplement: Bouillon fortified with FePP + Stabilizer
  Arms: FePP + Stabilizer
Dietary Supplement: Bouillon fortified with FeSO4
  Arms: FeSO4
Dietary Supplement: Bouillon fortified with FeSO4 + Stabilizer
  Arms: FeSO4 + Stabilizer

SUMMARY:
Iron deficiency is a highly prevalent nutrient deficiency which is a public health problem, especially in developing countries. There are several strategies to correct iron deficiency in populations: besides supplementation with tablets, one of the most sustainable and effective strategies on medium term has been iron fortification, the addition of iron to regularly consumed foods. In fortification, the chemical nature of the compound to be added plays an important role: depending on the compound sensory qualities of the fortified foods can vary as well as the iron absorption. Iron pyrophosphate (FePP) and ferrous sulfate (FeSO4) are two commonly used iron fortification compounds in foods such as rice, breakfast cereals, pasta, flour and others. We want to test the effect of addition a food stabilizer on the absorption of ferric pyrophosphate (FePP) and ferrous sulfate (FeSO4) when added to bouillon, as was recently suggested by in vitro experiments in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 40 years at screening;
* Body weight <65 kg;
* Apparently healthy: no medical conditions which might affect study measurements (judged by study physician);
* With low iron stores (serum ferritin <15µg/L);
* Reported intense sporting activities ≤10h/w;
* Reported alcohol consumption ≤14 units/w;
* Currently not smoking and being a non-smoker for at least six months and no reported use of any nicotine containing products in the six months preceding the study and during the study itself;
* Willing and able to participate in the study;
* Having given a written informed consent.

Exclusion Criteria:

* Being an employee of Unilever or the Laboratory of Human Nutrition of the ETH Zürich;
* Blood donation or significant blood loss over the past 6 months;
* Reported use of any medically- or self-prescribed diet;
* Use of medication (except oral contraceptives)
* Use of vitamin or mineral supplements and unwillingness to discontinue their use two weeks prior the study and during the study;
* Smoking or consuming tobacco in any form, and/or was smoking or consuming tobacco in any form for 6 months preceding the study and/or will be smoking or consuming tobacco in any form, during the study;
* Is pregnant or will be planning pregnancy during the study period;
* Is lactating or has been lactating in the 6 weeks before pre-study investigation and/or during the study period;
* Known gastrointestinal or metabolic disorders;
* Moderate or severe anemia defined as Hb < 90 g/L.
* Participation in another clinical trial during the last 30 days prior to the beginning of the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 2 | baseline, 2 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 4 in the isotopic ratio of iron in blood at week 6 | 4 weeks, 6 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.